CLINICAL TRIAL: NCT00884754
Title: Comparison of GlideScope-Specific Rigid Stylet to Standard Malleable Stylet for GlideScope Intubation by Novice Operators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Philip Jones, University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: R-08-594; 15520 (Other: REB)
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-12

CONDITIONS: Airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rigid GlideScope Specific Stylet (Experimental)
  Interventions: Device: GlideScope rigid stylet
- 90º curvature, malleable stylet (Active Comparator)
  Interventions: Device: GlideScope rigid stylet

INTERVENTIONS:
Device: GlideScope rigid stylet — Patients will be intubated either with a rigid stylet meant to be used with the GlideScope, or with a standard malleable stylet used with other modalities of intubation.

SUMMARY:
Patients presenting for elective surgery requiring tracheal intubation will be randomized to one of two different endotracheal tube (ETT) stylets. The intubation will be done with a GlideScope videolaryngoscope by a novice operator. The primary outcome is time to intubation.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient scheduled for elective surgery.
* ETT is indicated for the procedure in the opinion of the attending anesthesiologist.
* any operator who has performed ≤ 10 GlideScope intubations.

Exclusion Criteria:

* any patient in whom the use of the GlideScope is contraindicated in the opinion of the attending anesthesiologist.
* Patient with known cervical spine abnormalities.
* any patients with known or probable difficult airways. (This rare occurrence is unlikely to be evenly distributed between the groups and could skew the data).
* any patient requiring rapid sequence induction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jones, MD, FRCPC, Principal Investigator — LHSC
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Jones PM, Loh FL, Youssef HN, Turkstra TP. A randomized comparison of the GlideRite((R)) Rigid Stylet to a malleable stylet for orotracheal intubation by novices using the GlideScope((R)). Can J Anaesth. 2011 Mar;58(3):256-61. doi: 10.1007/s12630-010-9440-z. Epub 2010 Dec 17. PMID 21165728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rigid GlideScope Specific Stylet | 90º Curvature, Malleable Stylet
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rigid GlideScope Specific Stylet | 90º Curvature, Malleable Stylet | Total
Number analyzed (Participants) | 30 | 30 | 60
Age Categorical [Number; unit: participants]
  Over 18 years | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation (Seconds)
Time Frame: 30-150 seconds (anticipated)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Rigid GlideScope Specific Stylet | 90º Curvature, Malleable Stylet
Number analyzed (Participants) | 30 | 30
seconds | 60 [48 to 75] | 61 [49 to 75]

ADVERSE EVENTS:
Arm/Group | Rigid GlideScope Specific Stylet | 90º Curvature, Malleable Stylet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No